CLINICAL TRIAL: NCT01032785
Title: Timing of Closure of Patent Foramen Ovale and Patent Ductus Arteriosus Following Birth
Brief Title: Timing of Closure of Patent Foramen Ovale Following Birth
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Wolfson Medical Center (Other Government)
Responsible Party: Dr. Akiva Tamir, Head of Pediatric Cardiology Unit
Other Study IDs: 0049-09-WOMC
Record Dates: First submitted 2009-12-15; First posted 2009-12-16 (Estimated); Last update posted 2010-09-14 (Estimated); Status verified 2010-09

CONDITIONS: Closure of the Foramen Ovale and Ductus Arteriosus
Keywords: Patent Foramen Ovale; Patent Ductus Arteriosus; PFO; PDA
MeSH Terms: conditions — Ductus Arteriosus, Patent; Foramen Ovale, Patent

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Healthy term newborn: Any healthy term newborn born in Wolfson Medical Center
  Interventions: Device: no interventions

INTERVENTIONS:
Device: no interventions — no interventions

SUMMARY:
It is known that the foramen ovale closes in most infants during the first 6 months of life, however, most of the important papers in the field concentrated on observing infants with murmurs and following those with patent foramen ovale by echocardiography until 6-24 months. The purpose of this study is to observe the natural profile of closure of the foramen ovale and ductus arteriosus for the first 36 hours after birth. This understanding may help to avoid unnecessary treatment and exams for newborns with findings that are natural for their stage of development.

DETAILED DESCRIPTION:
We will observe the patency and size of foramen ovale five times within the first 36 hours of life. We will also describe the anatomy of the foramen ovale and the septum primum during this time. The direction of flow across the foramen ovale will also be observed. Other cardiac lesions will be checked for as well. We will measure the change in size of the pulmonary arteries and the closure of the ductus arteriosus.

ELIGIBILITY:
Inclusion Criteria:

* any baby born in term and with normal delivery

Exclusion Criteria:

* sick newborns in need of neonatal intensive care for any medical reason.
* newborns with congenital heart disease except for small, muscular ventricular septal defects

Ages: 30 Minutes to 4 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Population consits of newborn babies born in term and under normal delivery in Wolfson M.C.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2009-12; Primary Completion 2010-03 (Estimated); Study Completion 2010-03 (Estimated)

PRIMARY OUTCOMES:
Patent Foramen Ovale size using 2 echocardiography positions, shunt direction and distance of septum primum to Superior Vena Cava | 2-3 hours after birth, 5-6 hours, 7-8 hours, 12-13 hours and 36 hours

SECONDARY OUTCOMES:
Patent Ductus Arteriosus size, shunt direction and the size of the Left Pulmonary Artery, the Right Pulmonary Artery and the Pulmonary Annulus | 2-3 hours after birth, 5-6 hours, 7-8 hours, 12-13 hours, 36 hours

CONTACTS AND LOCATIONS:
Overall Officials: Akiva Tamir, M.D, Principal Investigator — Tel Aviv University
Locations (1):
- Wolfson Medical Center, Holon, Israel